CLINICAL TRIAL: NCT04242576
Title: Evaluation of Nociceptive Processing in the Cervical Region Through Action Observation, Laterality Discrimination and Exercise
Brief Title: Evaluation of Nociceptive Processing in the Cervical Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Josue Fernandez Carnero (Other)
Collaborators: Centro Universitario La Salle (Other)
Responsible Party: Sponsor-Investigator, Josue Fernandez Carnero, Professor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: URJC-07/2019
Record Dates: First submitted 2019-12-20; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Pain, Neck
Keywords: Neck; Graded motor imagery; Exercise; Action Observation; Right/Left judgment tasks
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Action Observation (Experimental): Subjects will watch 30-second videos, with a one-minute break between videos. The videos show the actions that subjects should imagine while watching the video.
  Interventions: Other: Action Observation
- Right/Left Judgment Task (Experimental): The laterality will be trained with the Recognize® application. Once the subjects have been trained, they are instructed to solve the different sections of the application, starting with the simplest tasks until reaching the most difficult ones.
  These tasks would consist of indicating "left" or "right", among the different images that appear on the iPad screen, indicating if the image's neck is rotated to the left or right. Being every level more complicated, so that people of different skin tones, with clothes or in a work environment are added.
  Interventions: Device: Right Left Judgement
- Exercise (Active Comparator): The subjects perform the exercises provided by the researchers. Which consist of neck exercises in all ranges of movement (inclinations and rotations to both sides), apart from flexion and extension.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Device: Right Left Judgement — It is an application by Noigroup (Neuro Orthopedic Institute), adapted to different devices.
  Other Names: Recognise® by Noigroup
  Arms: Right/Left Judgment Task
Other: Action Observation — Videos of cervical movements.
  Arms: Action Observation
Behavioral: Exercise — Evidence based exercises for the neck.
  Arms: Exercise

SUMMARY:
The main objective of this research is to asses the effectivity of action observation therapy, left/right discrimination and therapeutic exercise in the nociceptive processing of the cervical region.

DETAILED DESCRIPTION:
Neck pain is the fourth cause of loss of years due to disability, behind back pain, depression and joint pain. Studies show that about half of the population will experience at least one episode of the clinically important neck during their life. The vast majority of studies indicate a prevalence of neck pain that varies between 15% and 50%, including a systematic review with a ratio of 37.2%, the investigators can ensure that neck pain is a common pathology among the population. Among the variables associated with neck pain, besides rheumatology, include genetic, psychopathological variables (such as depression, anxiety, coping skills, somatization), sleep disorders, smoking and a sedentary lifestyle, among others. All those variables alter the nervous system in a proprioceptive level, so that deep and superficial flexor, as well as the rest of the muscles, they do not receive correct information that prevents them from processing properly the obtained information. Therefore, alterations also occur at central nervous system levels as in the processing of pain and its control by inhibitory descending systems.

The most used treatment for neck pain is exercise. In a recent Cochrane review conducted by Gross A. et al., It has been proven, despite the shortage of high-quality studies, that the use of exercise routines based on strength and resistance training causes a reduction in pain.

Motor imagery (MI) or graduated motor imagery (GMI) is defined as "the mental and dynamic process of action, without real movement execution" and the action observation (AO) consists in observing an action carried out by another person. These treatments are based on the ability of the nervous system to assimilate the images seen and process them until they reach the motor cortex, and thanks to the mirror neurons, the painful pattern decreases until it disappears. Thus, visualising a painful situation provokes and evokes in the brain, a painful experience, even when this is not actually happening.

Therefore, the interruption of this neural network of cortical proprioceptive representations and integration of motor processes, also known as "body schema", is particularly relevant for movement and manual therapies. One way to measure the current state of the body scheme is through laterality tasks or "left / right judgement task" (LRJT), which have proven to be an effective and reliable tool and can also be used as a treatment.

All of the above facilitates the possibility of using these tools as treatments focused on the cortical area with GMI. However, the effectiveness of MI is controversial. Some studies have been carried out in pathological patients, in a pilot study they confirmed the changes produced in the neck region, both by an increase in the range of movement and an increase in the pain threshold to pressure, focused on the population with chronic neck pain. It is difficult to find studies in healthy patients, although in recent years some publications on motor imagery can be found finding changes in the descending inhibitory systems of pain and its processing. Many variables such as the duration of the sessions, the time per exercise or the type of tasks to be performed, together with the lack of studies on the neck region and the comparison between different tasks and their respective affectation of the descending pain inhibitory systems, have led us to carry out this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers.
* Asymptomatic on cervical region.
* Understands and accept the informed consent.
* Spanish speakers.
* People with no cognitive disorders.

Exclusion Criteria:

* Pregnant women.
* Positive neurological signs or evidence of spinal cord compression (abnormal diffuse sensitivity, hyperreflexia or diffuse weakness).
* Previous cervical surgeries with recurrent symptoms.
* Previous headaches.
* Inability to provide informed consent.
* Cognitive disorders.
* Reading or verbal misunderstanding when receiving instructions.
* Having suffered any pain in the last 3 months, both in the quadrant suppressor as in the lumbar region and pelvis.
* Suffer any pain at the time of the study.
* Any recent traumatic event, whether physical or psychological / emotional.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in cervical range of movement. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  Measured with goniometer by the physiotherapists.
Changes in pain perception. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  Self reported Visual Analog Scale. Minimum value is 0 (best); Maximun value is 10 (worst).
Changes in the subject's selective attention capacity and skills as well as their processing speed ability. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  It will be measured using the Encephalapp application. The time taken to perform 2 successful trials of 10 images without making an error was recorded.
Changes in pain treshold perception. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  Mechanical nociceptive threshold test using Von-Frey filaments.
Changes in upper Limb Neurodinamics. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  Upper limb neurodinamics test measuring with a goniometer on what grade of joint movement with nerve stretching pain appears.
Changes in levels of hyperalgesia to pressure and maximum pressure tolerance. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  Pressure Pain Tresholds using an algometer on first finger, trapezius muscle and tibia.
Changes in endogenous pain inhibition mechanisms. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  Conditioned pain modulation and temporal summation (windup), using the algometer and an oclussion band.
Changes in pain to cold threshold. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  Cold stimulation test using cold compresses on the cervical region two times during 10 minutes.
Changes in deep neck flexors activation. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  Deep neck flexor endurance test.
Changes in hand and forearm muscular strenght. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  Handgrip strenght test using a dynamometer.

SECONDARY OUTCOMES:
Changes in levels of Catastrophism. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  13 item Pain Catastrophic Scale that must be answered with a numeric value between 0 (not at all) and 4 (all the time), with a maximum score of 52 points, with higher scores indicating greater pain catastrophizing.
Changes in Kinesiophobia, levels of fear to movement. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  11 item Tampa Scale for Kinesiophobia, the final score can range between 11 and 44 points, with higher scores indicating greater perceived kinesiophobia.
Changes in Fear-avoidance behaviours. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  Fear-avoidance Beliefs Questionnaire . The instrument consists of two subscales, a four-item physical activity subscale, and a seven-item work subscale. Each item is scored from 0 to 6 and summed to produce the subscale score. Possible scores range from 0-28 to 0-42, with higher scores indicating greater fear avoidance beliefs.
Changes in level of Depression. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  Beck's Depression Inventory II is a 21-item self-reporting questionnaire. It scores from 0 to 21, the higher is the score the higher is the level of depression.
Changes in patient's anxiety. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  State-Trait Anxiety Inventory. The total score ranges from 0-63 interpreted as follows: 0-9, normal or no anxiety; 10-18, mild to moderate anxiety; 19-29, moderate to severe anxiety; and 30-63, severe anxiety.
Changes in the ability to generate mental motor images. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  The Movement Imagery Questionnaire-Revised. It is an 8-item self-reporting inventory rating the difficulty of generating that image on a 7-point scale, where 1 indicates 'very difficult to see/feel' and 7 indicates 'very easy to see/feel'.

OTHER OUTCOMES:
Physical activity of the patients. | Before and after the treatment (2 weeks), after 15 days and after 30 days.
  International physical activity questionnaire. Results are reported in categories depending on the variable 'MET minutes a week'. MET minutes represent the amount of energy expended carrying out physical activity. High physical activity (one hour of more of physical activity per day), moderate physical activity (half an hour of physical activity per day) or low physical activity (not meeting any of the criteria for either moderate or high levels of physical activity).

CONTACTS AND LOCATIONS:
Overall Officials: David Morales Tejera, Msc., Phdc, Principal Investigator — Universidad Rey Juan Carlos
Locations (2):
- Spain (2):
  - Centro superior de Estudios Universitarios La Salle, Madrid, Aravaca
  - Universidad Rey Juan Carlos, Alcorcón, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murray CJ, Atkinson C, Bhalla K, Birbeck G, Burstein R, Chou D, Dellavalle R, Danaei G, Ezzati M, Fahimi A, Flaxman D, Foreman, Gabriel S, Gakidou E, Kassebaum N, Khatibzadeh S, Lim S, Lipshultz SE, London S, Lopez, MacIntyre MF, Mokdad AH, Moran A, Moran AE, Mozaffarian D, Murphy T, Naghavi M, Pope C, Roberts T, Salomon J, Schwebel DC, Shahraz S, Sleet DA, Murray, Abraham J, Ali MK, Atkinson C, Bartels DH, Bhalla K, Birbeck G, Burstein R, Chen H, Criqui MH, Dahodwala, Jarlais, Ding EL, Dorsey ER, Ebel BE, Ezzati M, Fahami, Flaxman S, Flaxman AD, Gonzalez-Medina D, Grant B, Hagan H, Hoffman H, Kassebaum N, Khatibzadeh S, Leasher JL, Lin J, Lipshultz SE, Lozano R, Lu Y, Mallinger L, McDermott MM, Micha R, Miller TR, Mokdad AA, Mokdad AH, Mozaffarian D, Naghavi M, Narayan KM, Omer SB, Pelizzari PM, Phillips D, Ranganathan D, Rivara FP, Roberts T, Sampson U, Sanman E, Sapkota A, Schwebel DC, Sharaz S, Shivakoti R, Singh GM, Singh D, Tavakkoli M, Towbin JA, Wilkinson JD, Zabetian A, Murray, Abraham J, Ali MK, Alvardo M, Atkinson C, Baddour LM, Benjamin EJ, Bhalla K, Birbeck G, Bolliger I, Burstein R, Carnahan E, Chou D, Chugh SS, Cohen A, Colson KE, Cooper LT, Couser W, Criqui MH, Dabhadkar KC, Dellavalle RP, Jarlais, Dicker D, Dorsey ER, Duber H, Ebel BE, Engell RE, Ezzati M, Felson DT, Finucane MM, Flaxman S, Flaxman AD, Fleming T, Foreman, Forouzanfar MH, Freedman G, Freeman MK, Gakidou E, Gillum RF, Gonzalez-Medina D, Gosselin R, Gutierrez HR, Hagan H, Havmoeller R, Hoffman H, Jacobsen KH, James SL, Jasrasaria R, Jayarman S, Johns N, Kassebaum N, Khatibzadeh S, Lan Q, Leasher JL, Lim S, Lipshultz SE, London S, Lopez, Lozano R, Lu Y, Mallinger L, Meltzer M, Mensah GA, Michaud C, Miller TR, Mock C, Moffitt TE, Mokdad AA, Mokdad AH, Moran A, Naghavi M, Narayan KM, Nelson RG, Olives C, Omer SB, Ortblad K, Ostro B, Pelizzari PM, Phillips D, Raju M, Razavi H, Ritz B, Roberts T, Sacco RL, Salomon J, Sampson U, Schwebel DC, Shahraz S, Shibuya K, Silberberg D, Singh JA, Steenland K, Taylor JA, Thurston GD, Vavilala MS, Vos T, Wagner GR, Weinstock MA, Weisskopf MG, Wulf S, Murray; U.S. Burden of Disease Collaborators. The state of US health, 1990-2010: burden of diseases, injuries, and risk factors. JAMA. 2013 Aug 14;310(6):591-608. doi: 10.1001/jama.2013.13805. PMID 23842577
- [Background] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284
- [Background] Cohen SP. Epidemiology, diagnosis, and treatment of neck pain. Mayo Clin Proc. 2015 Feb;90(2):284-99. doi: 10.1016/j.mayocp.2014.09.008. PMID 25659245
- [Background] Falla D, Jull G, Russell T, Vicenzino B, Hodges P. Effect of neck exercise on sitting posture in patients with chronic neck pain. Phys Ther. 2007 Apr;87(4):408-17. doi: 10.2522/ptj.20060009. Epub 2007 Mar 6. PMID 17341512
- [Background] Cohen SP, Hooten WM. Advances in the diagnosis and management of neck pain. BMJ. 2017 Aug 14;358:j3221. doi: 10.1136/bmj.j3221. PMID 28807894
- [Background] Kay TM, Gross A, Goldsmith CH, Rutherford S, Voth S, Hoving JL, Bronfort G, Santaguida PL. Exercises for mechanical neck disorders. Cochrane Database Syst Rev. 2012 Aug 15;(8):CD004250. doi: 10.1002/14651858.CD004250.pub4. PMID 22895940
- [Background] Losana-Ferrer A, Manzanas-Lopez S, Cuenca-Martinez F, Paris-Alemany A, La Touche R. Effects of motor imagery and action observation on hand grip strength, electromyographic activity and intramuscular oxygenation in the hand gripping gesture: A randomized controlled trial. Hum Mov Sci. 2018 Apr;58:119-131. doi: 10.1016/j.humov.2018.01.011. Epub 2018 Mar 12. PMID 29408163
- [Background] La Touche R, Grande-Alonso M, Cuenca-Martinez F, Gonzalez-Ferrero L, Suso-Marti L, Paris-Alemany A. Diminished Kinesthetic and Visual Motor Imagery Ability in Adults With Chronic Low Back Pain. PM R. 2019 Mar;11(3):227-235. doi: 10.1016/j.pmrj.2018.05.025. Epub 2019 Jan 15. PMID 29908933
- [Background] Schmid AB, Coppieters MW. Left/right judgment of body parts is selectively impaired in patients with unilateral carpal tunnel syndrome. Clin J Pain. 2012 Sep;28(7):615-22. doi: 10.1097/AJP.0b013e31823e16b9. PMID 22688599
- [Background] Wallwork SB, Butler DS, Fulton I, Stewart H, Darmawan I, Moseley GL. Left/right neck rotation judgments are affected by age, gender, handedness and image rotation. Man Ther. 2013 Jun;18(3):225-30. doi: 10.1016/j.math.2012.10.006. Epub 2013 Jan 26. PMID 23357411